CLINICAL TRIAL: NCT02181621
Title: A Prospective, Open, Comparative, Randomized, Single-centre Study to Evaluate the Effect of Cadexomer Iodine Gel (IODOSORB) Compared to Standard Dressings (SOLOSITE) on Biofilm Disruption in Infected Diabetic Foot Ulcers (DFUs)
Brief Title: A RCT to Compare the Effects of Two Wound Products on Biofilm Disruption in DFUs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE048IOD
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2015-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solosite gel (Placebo Comparator): Hydrogel with preservatives, used to create a moist wound environment.
  Interventions: Device: Solosite gel
- Iodosorb (Active Comparator): Cadexomer iodine gel
  Interventions: Device: Iodosorb

INTERVENTIONS:
Device: Iodosorb — Cadexomer iodine gel
  Arms: Iodosorb
Device: Solosite gel — Hydrogel
  Arms: Solosite gel

SUMMARY:
This study is a prospective comparative study to determine if an Iodine Gel (Iodosorb◊) is better than standard dressing (Solosite◊ gel) in disruption of biofilm (small microorganism bacteria similar to plaque on teeth) on the wound bed diabetic foot ulcers.

◊ Trademark of Smith & Nephew

DETAILED DESCRIPTION:
IODOSORB gel is a cadexomer iodine product indicated for use in wet ulcers and wounds. As the use of IODOSORB has an anti-microbial effect and removes exudate continuously from the wound, a reduction in pain, odour, oedema, exudate, pus and debris, and microbial load including biofilm can be achieved, hence providing an environment conducive to the normal healing process. While evidence exists to support the use of IODOSORB in diabetic foot ulcers (DFUs) for the reduction of planktonic bacteria, little evidence exits for the effect of any topical therapy on non-planktonic or biofilm bacteria in-vivo. The aim of this study is to explore the effects of IODOSORB on biofilm in the wound, wound healing, and associated factors, such as odour, pain, and reduction of slough.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is able to understand the study and is willing to consent to the study.
2. The patient consents to the ongoing use of their de-identified photos by the Sponsor for purposes outside of this study.
3. The patient must be at least 18 years of age.
4. Males and females - provided they are not pregnant or lactating and if of reproductive age are using contraception.
5. The patient has presented with a DFU which, according to the clinical judgement of the Investigator, has a suspected biofilm
6. The patient has a DFU of Grade 1 or 2 according to the Meggit-Wagner scale. Grade 1 - Superficial ulcers limited to the dermis Grade 2 - Ulcers are transdermal with exposed bone or tendon, and without osteomyelitis or abscess formation
7. The patient's ulcer is suitable to be dressed with IODOSORB or SOLOSITE.
8. The patient has an ABPI >0.49; or toe pressure >50mmHg.

Exclusion Criteria:

1. Patients with a known history of poor compliance with medical treatment.
2. Patients who have participated in this study previously and who healed or were withdrawn.
3. Patients who are participating in any other clinical study.
4. Patients that have received continuous treatment with Iodosorb (on any wound) in the past 8 weeks (Iodosorb must not be continuously used for more 3 months) or whose reference ulcer has been treated with Iodosorb in the past 2 weeks.
5. Patients with a history of any thyroid disorders, e.g. Hashimoto's thyroiditis, Graves disease or non-toxic nodular goitre.
6. Patients undergoing treatment with mercurial antiseptics, taurolidine or lithium.
7. Patients with a known sensitivity to iodine or any of the other ingredients in IODOSORB, SOLOSITE or ALLEVYN Non-adhesive
8. Patients with severe renal impairment
9. Patients with an ulcer less than 3cm diameter.
10. Patients with an ulcer that is not exuding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lantis, BSc, MD, Principal Investigator — St Lukes Roosevelt Hospital Center; Matthew Christensen, Study Chair — Smith & Nephew, Inc. - SVP Global Clinical & Medical Affairs
Locations (1):
- St Lukes Roosevelt Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial assessment screening/enrollment occurred at a single site in the United States from 05Aug2014 to 11Sep2015. Eligible participants were randomized to receive either IODOSORB or SOLOSITE for up to 4 weeks (28 +/- 4 days) or until reference ulcer closure (whichever came first).
Groups:
- SOLOSITE: Hydrogel with preservatives, used to create a moist wound environment.
  SOLOSITE Gel: Hydrogel
Period: Overall Study
Arm/Group | SOLOSITE | IODOSORB
Started (Started = Initial Assessment) | 9 | 10
Week 1 Assessment | 7 | 8
Week 2 Assessment | 6 | 8
Week 3 Assessment | 6 | 7
Week 4 Assessment | 6 | 7
Completed | 7 | 8
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Previously Enrolled | 0 | 1
Not completed — Enrollment Hold | 1 | 1

BASELINE CHARACTERISTICS:
Population: The reporting of baseline measures is based on the confirmed biofilm analysis set, defined as all subjects enrolled in the study and available for analysis for which the presence of biofilm was confirmed using curettage samples.
Groups:
- Total: Total of all reporting groups
Arm/Group | SOLOSITE Gel | IODOSORB | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.2) | 51.4 (9) | 57 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Height (centimeters [cm]) [Mean (Standard Deviation); unit: cm] | 178.9 (12.6) | 179.9 (9.9) | 179.4 (10.9)
Weight (kilograms [kg]) [Mean (Standard Deviation); unit: kg] | 91.9 (31.5) | 114.5 (37.8) | 103.2 (35.5)
Baseline Reference Ulcer: Area (centimeters squared [cm^2]) [Median (Full Range); unit: cm^2] | 9.4 [5.1 to 21.2] | 8.5 [2.1 to 13.0] | 9 [2.1 to 21.2]
Baseline Reference Ulcer: Depth (millimeters [mm]) [Median (Full Range); unit: mm] | 4 [0.7 to 20] | 2 [0.2 to 6] | 3 [0.2 to 20]
Reference Ulcer: Volume (centimeters cubed [cm^3]) [Median (Full Range); unit: cm^3] | 3.8 [0.8 to 15.8] | 1.7 [0 to 6.4] | 2.3 [0 to 15.8]

OUTCOME MEASURES:

1. Primary Outcome: Within-patient Change From Baseline in Log^10 Biofilm-protected Bacteria Count (Colony Forming Units [Cfu]/Gram[g])
Description: The primary variable was the within-patient change from Baseline in log^10 biofilm-protected bacteria count from Baseline (initial assessment) to Week 4, as measured by curettage.
Time Frame: Baseline to Week 4
Population: The reporting of this outcome measure is based on the confirmed biofilm analysis set, defined as all subjects admitted to the study and for which the presence of biofilm was confirmed using curettage samples. Week 4 data were included for a total of 12 subjects (SOLOSITE N= 6; IODOSORB N = 6) in the biofilm analysis set.
Measure: Median (95% Confidence Interval); unit: log^10 CFU/g
Arm/Group | Solosite Gel | Iodosorb
Number analyzed (Participants) | 6 | 6
log^10 CFU/g | 0.8 [-1.1 to 3.5] | 1.0 [-2.2 to 5.8]

2. Secondary Outcome: Ulcer Area Measurements at Each Study Visit
Description: Calculated overall median/range measurements of the reference ulcer area (cm^2) at each study visit as well as overall study completion ulcer area measurements were assessed for the Iodosorb and Solosite arms. The ulcer area was calculated as area = length x width x 0.785.
Time Frame: Baseline up through Week 4 +/- 4 days or End of Study Visit, up to 32 days
Population: The reporting of this outcome measure is based on the confirmed biofilm analysis set, defined as all subjects admitted to the study and for which the presence of biofilm was confirmed using curettage samples (Initial Visit: N=14; Week 1: N=14; Week 2: N=13; Week 3: N=12; Week 4: N=12; Study Completion: N=14).
Measure: Median (Full Range); unit: cm^2
Arm/Group | Solosite Gel | Iodosorb
Number analyzed (Participants) | 7 | 7
cm^2
  Baseline Ulcer Area Measurement | 9.4 [5.1 to 21.2] | 8.5 [2.1 to 13.0]
  Week 1 Ulcer Area Measurement | 9.4 [3.9 to 19.4] | 7.3 [1.2 to 12.1]
  Week 2 Ulcer Area Measurement: number analyzed (Participants) | 6 | 7
  Week 2 Ulcer Area Measurement | 8.1 [4.0 to 14.1] | 7.8 [0.9 to 11.2]
  Week 3 Ulcer Area Measurement: number analyzed (Participants) | 6 | 6
  Week 3 Ulcer Area Measurement | 8.0 [2.9 to 12.0] | 7.0 [0.8 to 10.4]
  Week 4 Ulcer Area Measurement: number analyzed (Participants) | 6 | 6
  Week 4 Ulcer Area Measurement | 6.1 [4.4 to 9.7] | 6.8 [0.8 to 11.5]
  Study Completion Ulcer Area Measurement | 5.5 [4.4 to 9.7] | 7.8 [0.8 to 11.5]

3. Secondary Outcome: Percentage (%) Change in Ulcer Area
Description: Overall percentage (%) of change in ulcer area from Baseline to final visit for the Iodosorb and Solosite arms.
Time Frame: Baseline up through Week 4 +/- 4 days or End of Study Visit, up to 32 days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SOLOSITE | IODOSORB
Number analyzed (Participants) | 7 | 7
percent change | 29.4 (23.1) | 24.8 (39.0)

4. Secondary Outcome: Ulcer Depth Measurements at Each Study Visit
Description: Calculated median/range measurements of the reference ulcer depth (mm) at each study visit as well as overall study completion ulcer depth measurements were assessed for the Iodosorb and Solosite arms. The ulcer depth as measured by inserting the cotton applicator into the deepest part of the ulcer and measuring from the tip of the applicator to the level of the skin surface.
Time Frame: Baseline up through Week 4 +/- 4 days or End of Study Visit, up to 32 days
Population: as for outcome 2
Measure: Median (Full Range); unit: mm
Arm/Group | Solosite Gel | Iodosorb
Number analyzed (Participants) | 7 | 7
mm
  Baseline Ulcer Depth Measurement | 4 [0.7 to 20] | 2 [0.2 to 6]
  Week 1 Ulcer Depth Measurement | 3 [0.2 to 30] | 2 [1 to 4]
  Week 2 Ulcer Depth Measurement: number analyzed (Participants) | 6 | 7
  Week 2 Ulcer Depth Measurement | 2.5 [2 to 28] | 2 [1 to 3]
  Week 3 Ulcer Depth Measurement: number analyzed (Participants) | 6 | 6
  Week 3 Ulcer Depth Measurement | 2 [1 to 30] | 1.5 [1 to 3]
  Week 4 Ulcer Depth Measurement: number analyzed (Participants) | 6 | 6
  Week 4 Ulcer Depth Measurement | 2.5 [1 to 5] | 1.5 [1 to 3]
  Study Completion Ulcer Depth Measurement | 3 [1 to 5] | 2 [1 to 3]

5. Secondary Outcome: Percentage (%) Change in Ulcer Depth
Description: Overall percentage (%) of change in ulcer depth from Baseline to final visit for the Iodosorb and Solosite arms.
Time Frame: Baseline up through Week 4 +/- 4 days or End of Study Visit, up to 32 days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SOLOSITE | IODOSORB
Number analyzed (Participants) | 7 | 7
percent change | -7.9 (143.8) | -38.1 (165.2)

6. Secondary Outcome: Ulcer Volume Measurements at Each Study Visit
Description: Calculated median/range measurements of the ulcer volume (cm^3) at each study visit as well as overall study completion ulcer volume measurements were assessed for the Iodosorb and Solosite arms. The ulcer volume was measured by calculating the length x width x depth of the ulcer.
Time Frame: Baseline up through Week 4 +/- 4 days or End of Study Visit, up to 32 days
Population: as for outcome 2
Measure: Median (Full Range); unit: cm^3
Arm/Group | Solosite Gel | Iodosorb
Number analyzed (Participants) | 7 | 7
cm^3
  Baseline Ulcer Volume Measurement | 3.8 [0.8 to 15.8] | 1.7 [0.0 to 6.4]
  Week 1 Ulcer Volume Measurement | 3.3 [0.2 to 34.3] | 0.9 [0.1 to 3.6]
  Week 2 Ulcer Volume Measurement: number analyzed (Participants) | 6 | 7
  Week 2 Ulcer Volume Measurement | 2.6 [0.8 to 19.4] | 1.3 [0.2 to 3.4]
  Week 3 Ulcer Volume Measurement: number analyzed (Participants) | 6 | 6
  Week 3 Ulcer Volume Measurement | 1.7 [0.6 to 22.8] | 1.1 [0.1 to 3.0]
  Week 4 Ulcer Volume Measurement: number analyzed (Participants) | 6 | 6
  Week 4 Ulcer Volume Measurement | 1.8 [0.5 to 2.9] | 1.1 [0.1 to 2.4]
  Study Completion Ulcer Volume Measurement | 1.6 [0.5 to 2.9] | 1.1 [0.1 to 2.4]

7. Secondary Outcome: Percentage (%) Change in Ulcer Volume
Description: Overall percentage (%) of change in ulcer volume from Baseline to final visit for the Iodosorb and Solosite arms.
Time Frame: Baseline up through Week 4 +/- 4 days or End of Study Visit, up to 32 days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SOLOSITE | IODOSORB
Number analyzed (Participants) | 7 | 7
percent change | 15.0 (119.1) | 21.5 (57.5)

8. Secondary Outcome: Presence of Biofilm by Clinical Judgment Versus Presence of Biofilm by Laboratory Test
Description: Assessment of subjects clinically judged to have biofilm present on the wound. The presumption of biofilm was determined on visual appearance to the Investigator and compared to microbial swab laboratory test confirmation. Biofilm is a microbial colony encased in a polysaccharide matrix which can become attached to a wound surface and prevent healing. Biofilm can appear as a shiny or slimy layer (clear to yellowish in appearance) on a wound bed.
Time Frame: Baseline, Week 2, Week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SOLOSITE | IODOSORB
Number analyzed (Participants) | 7 | 7
Participants
  Biofilm Present by Laboratory Test at Baseline: Yes | 7 | 7
  Biofilm Present by Laboratory Test at Baseline: No | 0 | 0
  Biofilm Present by Clinical Judgment at Baseline: Yes | 7 | 7
  Biofilm Present by Clinical Judgment at Baseline: No | 0 | 0
  Biofilm Present by Laboratory Test at Week 2: number analyzed (Participants) | 6 | 7
  Biofilm Present by Laboratory Test at Week 2: Yes | 6 | 6
  Biofilm Present by Laboratory Test at Week 2: No | 0 | 1
  Biofilm Present by Clinical Judgment at Week 2: number analyzed (Participants) | 6 | 7
  Biofilm Present by Clinical Judgment at Week 2: Yes | 6 | 5
  Biofilm Present by Clinical Judgment at Week 2: No | 0 | 2
  Biofilm Present by Laboratory Test at Week 4: number analyzed (Participants) | 6 | 6
  Biofilm Present by Laboratory Test at Week 4: Yes | 5 | 4
  Biofilm Present by Laboratory Test at Week 4: No | 1 | 2
  Biofilm Present by Clinical Judgment at Week 4: number analyzed (Participants) | 6 | 6
  Biofilm Present by Clinical Judgment at Week 4: Yes | 5 | 4
  Biofilm Present by Clinical Judgment at Week 4: No | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of randomization up through 28 days (+/- 4 days).
Arm/Group | Solosite Gel | Iodosorb
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10
Other Adverse Events (participants affected / at risk) | 1/9 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solosite Gel (N=9) | Iodosorb (N=10)
Right Foot Abscess with Osteomyelitis (General disorders) | 0 (0) | 1 (1) — Right foot abscess with osteomyelitis; right proximal phalanx and metatarsal head resection with washout and primary closure; not related to study or investigational product; resulted in study withdrawal.
Spinal Infection (General disorders) | 1 (1) | 0 (0) — Not related to study or investigational product; resulted in study withdrawal.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solosite Gel (N=9) | Iodosorb (N=10)
Foot Laceration (General disorders) | 1 (1) | 0 (0) — Patient visited emergency room due to having stepped on glass; not study or investigational product related.
Open Ulcer, Left Great Toe (General disorders) | 0 (0) | 1 (1) — Open ulcer (non-target ulcer) on left great toe which was not present one week prior; not related to study or investigational product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No